CLINICAL TRIAL: NCT02868320
Title: SMS Technology for the Promotion of Diabetes Education and Self-Management
Brief Title: SMS Technology for the Promotion of Diabetes Education and Self-Management in Egypt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Haitham Abaza, Doctoral candidate at PLRI Institute for Medical Informatics, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DiabAwPro
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
Keywords: SMS; text messaging; diabetes self management; glycemic control; mHealth; mobile health; diabetes education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention group (Experimental): This group received a diabetes instruction booklet in addition to daily educational SMS messages and weekly reminders
  Interventions: Other: SMS messages; Other: Instruction booklet
- Control group (Active Comparator): This group only received a diabetes instruction booklet
  Interventions: Other: Instruction booklet

INTERVENTIONS:
Other: SMS messages — Daily educational messages addressing the following categories: diet, exercise, complications, medications, foot care, blood sugar testing, and hypo- and hyperglycemia.
  Weekly reminder messages of blood glucose testing.
  Arms: Intervention group
Other: Instruction booklet — General detailed instructions addressing the same SMS categories.

SUMMARY:
This study was conducted at the teaching hospital of Misr University for Science & Technology. It aimed to examine the use of SMS technology in educating and monitoring diabetic patients in Egypt, and assess the impact of educational text messages on their glycemic control and self-management behaviors. Participants were randomized into an intervention and a control group. Intervention patients received an instruction booklet as well as daily educational and weekly reminder messages to better control their diabetes. Control patients received the same instruction booklet but no SMS messages. Both group patients took an HbA1c test at the beginning and end of the study period and were asked to measure their blood glucose once a week and record their readings into a monitoring table over 12 weeks. The primary outcome was the change in HbA1c levels, which was expected to be greater among intervention patients at the end of the study. Secondary outcomes included blood glucose levels, treatment and medication adherence, diabetes self-efficacy, rate of hospital/ER visits, frequency of blood glucose measurement, among others.

ELIGIBILITY:
Inclusion Criteria:

* has diabetes
* owns a mobile phone
* can read SMS messages or lives with someone that can read for them.

Exclusion Criteria:

* cannot read or not SMS familiar and lives alone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
change in HbA1c | baseline and 12 weeks
  measured by the difference between endpoint and baseline values and by the number of patients who experienced a reduction of at least 1% from baseline to endpoint

SECONDARY OUTCOMES:
blood glucose levels | 12 weeks
body weight | 12 weeks
Treatment adherence | 12 weeks
  measured by the diabetes self-care inventory (SCI)
Medication adherence | 12 weeks
  measured by the Morisky medication adherence scale (MMAS-4)
Diabetes self-efficacy | 12 weeks
  measured by the diabetes empowerment scale short form (DES-SF)
Frequency of blood glucose measurement | 12 weeks
Rate of hospital/ER admissions | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Abaza, Principal Investigator — PLRI Institute for Medical Informatics, Hannover Medical School; Michael Marschollek, Study Director — PLRI Institute for Medical Informatics, Hannover Medical School
Locations (1):
- Misr University for Science & Technology (MUST) hospital, Giza, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Abaza H, Marschollek M. SMS education for the promotion of diabetes self-management in low & middle income countries: a pilot randomized controlled trial in Egypt. BMC Public Health. 2017 Dec 19;17(1):962. doi: 10.1186/s12889-017-4973-5. PMID 29258499